CLINICAL TRIAL: NCT02104102
Title: Biomedical Instrumentation in the Study of Mirror Therapy in Elderly's Hands Motor Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Vale do Paraíba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 24581613.0.0000.5503
Record Dates: First submitted 2014-02-07; First posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-03

CONDITIONS: Muscle Weakness Conditions
Keywords: Elderly; mirror therapy; hands
MeSH Terms: interventions — Mirror Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirror group (Experimental): Composed of 30 volunteers who carry out the mirror therapy, whose name shall Mirror Group (MG).
  Interventions: Other: Mirror Therapy
- Control Group - kinesiotherapy (Experimental): Called by Control Group (CG), composed of 30 volunteers who will carry out the kinesiotherapy with the same sequence of movements for the Mirror Therapy that the MG, but without the view in the mirror, since it will be blocked.
  Interventions: Other: Kinesiotherapy

INTERVENTIONS:
Other: Mirror Therapy — Mirror Therapy, which is based on the activation of mirror neurons from the illusion generated by viewing the reflection of a member in a mirror, that is, intended to facilitate the movement through the practice of bilateral symmetric activities, since it is able to stimulate cortical plasticity, promoting reversal of the decrease and the reestablishment of motor function.
  Arms: Mirror group
Other: Kinesiotherapy — Hands movements.
  Arms: Control Group - kinesiotherapy

SUMMARY:
Check if the Mirror therapy represents an effective method in improving the motor activity of the hands of institutionalized elderly.

DETAILED DESCRIPTION:
Among the various functions impaired by aging there is the muscle function, which indirectly affects the quality of life for seniors, since it is crucial to the progressive increase of the debilitating condition, leading to difficulties in carrying out everyday tasks and often making them dependent on the assistance of others. The possible neural mechanisms underlying this decrease in muscle function associated with aging include changes undefined in Central Nervous System, a delay in conduction velocity of motor nerve fibers and in transmission of the neuromuscular junction. In this context, it is necessary to develop procedures that reduce the functional losses and decrease the negative effects of the aging process, increasing the quality of life for seniors. Mirror Therapy (MT) is the one of those possible procedures, which is based on the activation of mirror neurons from the illusion generated by viewing the reflection of a member in a mirror. When performing a movement with a member who is in your field of vision, generated the reflection in the mirror is able to offer the brain a new, albeit illusory visual stimulus, suggesting that covert member is moving. This illusion promotes the activation of mirror neurons located in the sensorimotor cortex region and the progression of therapy, this activation drives cortical plasticity that promotes the reestablishment of functions, such as motor coordination and increased range of motion. Therefore, MT is a promising technique to reduce the functional losses of aging. It is then suggested the implementation of a protocol for functional recovery of MT hands in institutionalized elderly and the measurement of electromyographic activity of the wrist, the range and speed of movement, the writing skill and the application of a questionnaire to Katz index calculation in order to investigate whether the technique can benefit this public.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old or more
* Institutionalized elderly
* Ability to understand and sign the Informed Consent Form. In case of illiteracy, the term will be read to the volunteer and signed by him in the case of functional illiteracy or by officials of the asylum
* Ability to perform analysis of writing skills throughout the proposed protocol
* Cognitive preserved, being able to respond to the examiner's command

Exclusion Criteria:

* Disabling pain to perform movements with their arms
* Active infection and rash at the application site of EMG
* Severe uncorrected visual deficit
* Deficit uncorrected severe hearing
* Neurological disorders

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-07 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Electromyography | 6 weeks
  Muscle electrical activity will be assessed at two different times, one related to the collection along with the dynamometer and another related to the simultaneous collection accelerometer.It is expected that after treatment with Mirror Therapy for 2 weeks has been an improvement of sensorimotor functions, gain muscle strength , uniformity of muscle fiber recruitment and improves muscle synergy and gain in speed of movements.
Dynamometry | 6 weeks
  Manual strength will be assessed with the electromyography, asking the volunteer to perform the maximal volunteer contraction when pressing the portable manual dynamometer. It is expected that after treatment with Mirror Therapy for 2 weeks has been an improvement of muscle strength.
Functionality | 6 weeks
  The functionality will be measure by the Katz index during the period of the study.

SECONDARY OUTCOMES:
Range of motion | 6 weeks
  The range of motion will be taken for the movements of flexion and extension of the wrist.
Writing skill | 6 weeks
  The volunteers will writing a specified phrase and they will received a paper with four four geometric forms (square, triangle, circle and rhombus) to follow the line. This task should be done for both hands. The skill will be analysed by using a computer software developed to calculate the distances between the original line of the form and the line performed by the volunteer.

CONTACTS AND LOCATIONS:
Overall Officials: Rani S Alves, Graduate, Principal Investigator — Universidade do Vale do Paraíba
Locations (1):
- Laboratory of Sensory and Motor Rehabilitation Engineering, São José dos Campos, São Paulo, Brazil